CLINICAL TRIAL: NCT06154252
Title: A Phase 1/2, Open-Label Study to Evaluate the Safety and Efficacy of Autologous CD19-specific Chimeric Antigen Receptor T Cells (CABA-201) in Subjects With Active Idiopathic Inflammatory Myopathy or Juvenile Idiopathic Inflammatory Myopathy
Brief Title: RESET-Myositis: An Open-Label Study to Evaluate the Safety and Efficacy of CABA-201 in Subjects With Active Idiopathic Inflammatory Myopathy or Juvenile Idiopathic Inflammatory Myopathy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cabaletta Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAB-201-002
Record Dates: First submitted 2023-11-16; First posted 2023-12-04 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Idiopathic Inflammatory Myopathy; Dermatomyositis; Anti-Synthetase Syndrome; Immune-Mediated Necrotizing Myopathy; Juvenile Dermatomyositis; Juvenile Polymyositis; Juvenile Idiopathic Inflammatory Myopathy (JIIM); Juvenile Myositis
Keywords: CABA-201; Autoimmune Disease; Anti-CD19 CAR-T therapy; Cellular Therapy; Idiopathic Inflammatory Myopathy; Myositis; Dermatomyositis; Anti-synthetase Syndrome; Immune-mediated Necrotizing Myopathy; Juvenile Dermatomyositis; Juvenile Polymyositis; Juvenile Idiopathic Inflammatory Myopathy (JIIM); Juvenile Myositis
MeSH Terms: conditions — Myositis; Dermatomyositis; Autoimmune Diseases | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CABA-201 (Experimental): DM Cohort: Infusion of CABA-201 following preconditioning with fludarabine and cyclophosphamide preconditioning in subjects with DM.
  ASyS Cohort: Infusion of CABA-201 following preconditioning with fludarabine and cyclophosphamide preconditioning in subjects with ASyS.
  IMNM Cohort: Infusion of CABA-201 following preconditioning with fludarabine and cyclophosphamide preconditioning in subjects with IMNM.
  JIIM Cohort: Infusion of CABA-201 following preconditioning with fludarabine and cyclophosphamide preconditioning in subjects with JIIM.
  Interventions: Biological: CABA-201 following preconditioning with fludarabine and cyclophosphamide

INTERVENTIONS:
Biological: CABA-201 following preconditioning with fludarabine and cyclophosphamide — Single intravenous infusion of CABA-201 at a single dose level following preconditioning with fludarabine and cyclophosphamide
  Other Names: Rese-cel; Resecabtagene autoleucel

SUMMARY:
RESET-Myositis: Open-Label Study to Evaluate the Safety and Efficacy of CABA-201 in Subjects with Active Idiopathic Inflammatory Myopathy or Juvenile Idiopathic Inflammatory Myopathy

DETAILED DESCRIPTION:
Idiopathic inflammatory myopathies (IIMs, or myositis) are a group of rare autoimmune diseases characterized by inflammation and muscle weakness. Though the cause of IIM is not well understood, some subtypes of IIM, including dermatomyositis (DM), anti-synthetase syndrome (ASyS), immune-mediated necrotizing myopathy (IMNM), and juvenile idiopathic inflammatory myopathy (JIIM), are thought to involve B cells that cause the body to attack different tissues in the body. This study is being conducted to evaluate the safety and efficacy of an investigational cell therapy, CABA-201, that can be given to patients with DM, ASyS, IMNM, or JIIM who have active disease. A single dose of CABA-201 in combination with cyclophosphamide (CY) and fludarabine (FLU) will be evaluated.

ELIGIBILITY:
Adult Cohorts

Inclusion Criteria:

* Age ≥18 and ≤75
* A clinical diagnosis of IIM, based on the 2017 The European League Against Rheumatism/American College of Rheumatology classification criteria
* Diagnosis of DM, ASyS, IMNM
* Evidence of active disease, despite prior or current treatment with standard of care treatments, as defined by the presence of elevated creatine kinase (CK), DM rash, or active disease on muscle biopsy, magnetic resonance imaging (MRI), or electromyography
* Presence of muscle weakness

Other protocol-defined criteria apply.

Exclusion Criteria:

* Contraindication to leukapheresis
* History of anaphylactic or severe systemic reaction to fludarabine, cyclophosphamide or any of their metabolites
* Active infection requiring medical intervention at screening
* Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, psychiatric, cardiac, neurological, or cerebral disease, including severe and uncontrolled infections, such as sepsis and opportunistic infections
* Concomitant medical conditions that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study, interfere with the assessment of the effects or safety of the investigational product or with the study procedures
* Significant lung or cardiac impairment
* Previous CAR T cell therapy
* Prior solid organ (heart, liver, kidney, lung) transplant or hematopoietic cell transplant

Other protocol-defined criteria apply.

Juvenile Cohort

Inclusion Criteria:

* Age ≥6 and ≤17 years at enrollment
* A clinical diagnosis of IIM, based on the 2017 The European League Against Rheumatism/American College of Rheumatology classification criteria
* Evidence of active disease, despite prior or current treatment with standard of care treatments, as defined by the presence of elevated muscle enzymes, DM rash, or active disease on muscle biopsy, magnetic resonance imaging (MRI), or electromyography

Other protocol-defined criteria apply.

Exclusion Criteria:

* Contraindication to leukapheresis
* History of anaphylactic or severe systemic reaction to fludarabine, cyclophosphamide or any of their metabolites
* Active infection requiring medical intervention at screening
* Current symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, pulmonary, psychiatric, cardiac, neurological, or cerebral disease, including severe and uncontrolled infections, such as sepsis and opportunistic infections.
* Concomitant medical conditions that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study, interfere with the assessment of the effects or safety of the investigational product or with the study procedures
* Significant lung or cardiac impairment
* Previous CAR T cell therapy
* Prior solid organ (heart, liver, kidney, lung) transplant or hematopoietic cell transplant

Other protocol-defined criteria apply.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate adverse events reported by subjects | Up to 28 days after CABA-201 infusion
  Incidence and severity of AEs

SECONDARY OUTCOMES:
To evaluate adverse events and laboratory abnormalities | Up to 156 weeks
  Incidence and severity of AEs, including changes in laboratory values and vital signs
To characterize the pharmacodynamics (PD) | Up to 156 weeks
  Levels of B cells in the blood
To characterize the pharmacokinetics (PK) | Up to 156 weeks
  Levels of CABA-201-positive T cells in the blood
To evaluate disease-related biomarkers of muscle inflammation | Up to 156 weeks
  Levels of muscle enzymes (CK, LDH, AST, ALT, and aldolase) in serum
To evaluate autoantibody -related biomarkers | Up to 156 weeks
  Levels of autoantibodies from the Myositis-Specific Autoantibody Panel (e.g., MDA-5, Jo-1, and HMGCR) in the serum
To evaluate efficacy | Up to 156 weeks
  Total Improvement Score (0 to 100, with higher scores indicating greater improvement) based on the Core Set Measures

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Cabaletta Bio
Locations (25):
- United States (21):
  - University of California Irvine - Accepting Adult Patients, Orange, California
  - University of California, San Francisco Benioff Children's Hospital - Accepting Young Adult and Juvenile Patients, San Francisco, California
  - Children's Hospital Colorado - Accepting Juvenile Patients, Aurora, Colorado
  - Mayo Clinic Florida - Accepting Adult Patients, Jacksonville, Florida
  - Emory University - Accepting Adult Patients, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago - Accepting Young Adult and Juvenile Patients, Chicago, Illinois
  - Northwestern Memorial Hospital - Accepting Adult Patients, Chicago, Illinois
  - The University of Chicago Medical Center - Accepting Adult and Juvenile Patients, Chicago, Illinois
  - University of Kansas Medical Center - Accepting Adult Patients, Kansas City, Kansas
  - National Institutes of Health - Accepting Adult and Juvenile Patients, Bethesda, Maryland
  - University of Michigan - Accepting Young Adult and Juvenile Patients, Ann Arbor, Michigan
  - Mayo Clinic - Accepting Adult Patients, Rochester, Minnesota
  - Hospital for Special Surgery - Accepting Adult and Juvenile Patients, New York, New York
  - Memorial Sloan Kettering Cancer Center - Accepting Adult and Juvenile Patients, New York, New York
  - Children's Hospital at Montefiore - Accepting Juvenile Patients, The Bronx, New York
  - Oregon Health & Science University - Accepting Adult Patients, Portland, Oregon
  - Children's Hospital of Philadelphia - Accepting Young Adult and Juvenile Patients, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center - Accepting Adult Patients, Nashville, Tennessee
  - Houston Methodist Hospital - Accepting Adult Patients, Houston, Texas
  - University of Texas MD Anderson Cancer Center - Accepting Adult Patients, Houston, Texas
  - Seattle Children's Research Institute - Accepting Juvenile Patients, Seattle, Washington
- United Kingdom (4):
  - Kings College Hospital NHS Foundation Trust - Accepting Adult Patients, London
  - University College London Hospitals NHS Foundation Trust - Accepting Adult Patients, London
  - Manchester Royal Infirmary - Accepting Adult Patients, Manchester
  - Salford Royal Hospital - Accepting Adult Patients, Salford

IPD SHARING:
Plan to Share IPD: No